CLINICAL TRIAL: NCT00889018
Title: Randomized Control Trial Comparing Carboplatin 560mg/m2 With 750mg/m2 for Ocular Salvage in Groups C and D Intraocular Retinoblastoma
Brief Title: Trial Comparing Two Carboplatin Doses in Groups C and D Intraocular Retinoblastoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: Council of Scientific and Industrial Research, India (Other Government)
Responsible Party: Principal Investigator, Rachna Meel, Senior Research Associate, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RACHNAMEEL
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Intraocular Retinoblastoma
Keywords: intraocular retinoblastoma; chemotherapy
MeSH Terms: interventions — Carboplatin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- group 1 (Active Comparator): chemotherapy using carboplatin 560mg/m2
  Interventions: Drug: carboplatin
- group 2 (Experimental): chemotherapy using 750mg/m2 carboplatin
  Interventions: Drug: carboplatin

INTERVENTIONS:
Drug: carboplatin — Table. 1: Chemotherapy protocol Vincristine Etoposide Carboplatin Day1 + + + Day2 ---- + ---- This regimen is repeated once a month for 6 months.Dose:Vincristine: 1.5 mg/m2 (0.05 mg/kg for children £36 months old and maximum dose 2 mg).Etoposide: 150 mg/m2 (5 mg/kg for children £36 months old).Carboplatin: 560 mg/m2 (18.6 mg/kg for children £36 months old). .
  Other Names: paraplatin
  Arms: group 1
Drug: carboplatin — Table. 1: Chemotherapy protocol Vincristine Etoposide Carboplatin Day1 + + + Day2 ---- + ---- This regimen is repeated once a month for 6 months.Dose:Vincristine: 1.5 mg/m2 (0.05 mg/kg for children £36 months old and maximum dose 2 mg).Etoposide: 150 mg/m2 (5 mg/kg for children £36 months old).Carboplatin: 750 mg/m2 (25 mg/kg for children £36 months old).
  Other Names: paraplatin
  Arms: group 2

SUMMARY:
The purpose of this study is to determine whether an increase in the dose of carboplatin in treatment of advanced intraocular (group C and D) retinoblastoma helps in avoiding radiotherapy and improves the rate of globe salvage.

DETAILED DESCRIPTION:
Chemoreduction has become an important method in management of retinoblastoma. This technique has been employed in an effort to avoid enucleation and external beam radiotherapy (EBRT) for children with intraocular retinoblastoma, especially those with bilateral disease. Although an ideal regimen for chemoreduction has not been determined, most authors use a combination of vincristine, etoposide and carboplatin for 2- 6 cycles along with local treatment including cryotherapy, laser photocoagulation, thermotherapy and plaque radiotherapy. Chemoreduction along with local treatment has been shown to have high treatment success in groups A and B of retinoblastoma allowing globe salvage without need of EBRT. But globe salvage rates remain low in groups C and D, which mostly need enucleation, or EBRT in a large number of cases.

In bilateral retinoblastoma where one eye is already lost owing to enucleation or both the eyes have advanced retinoblastoma (group C/D) globe salvage assumes a significant role in the overall treatment. Recurrences of the vitreous seeds or the sub retinal seeds are the main causes of treatment failure with chemoreduction and local treatment, ultimately requiring enucleation or EBRT.

The recurrence of vitreous or subretinal seeds do not necessarily mean a tumor resistance, it may reflect an inadequate penetration of the chemotherapeutic agents in these relatively avascular sites i.e the vitreous cavity or the subretinal space.

The penetration to these sites could be enhanced by (a) increase in the dose of the intravenous chemotherapeutic agents. The IInd Toronto protocol that was started in 2000 explores this option. The initial reports are encouraging but they have used high doses chemotherapy in combination with cyclosporin A. Therefore the effect of high dose chemotherapy on the globe salvage rates in groups C and D cannot be evaluated as an independent factor. (b) Periocular carboplatin injection has proven to deliver much higher levels of the drug in to the vitreous cavity, but several studies have revealed local side effects of this apparently harmless technique.The National Collaborative Retinoblastoma Study funded by the Children's oncology group plans to carry out a single arm trial of 6 cycles of systemic high dose chemotherapy and subtenon carboplatin injections in groups C and D of retinoblastoma. (c) Use of Cryotherapy/thermotherapy along with chemotherapy, has shown to increase the penetration of the chemotherapeutic agents into the vitreous cavity probably by disrupting the blood retinal barrier.

Shield's et al has already shown that the 6 cycle chemotherapy regimen achieves better long-term control of vitreous and subretinal seeds as compared to a 2 cycle regimen.

We planned this study to compare two different dose schedules of carboplatin and compare the rate of globe salvage in group C and D retinoblastoma and also to evaluate the effect of subtenon Carboplatin injections in cases that fail to respond to primary chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* All new cases of retinoblastoma with group C or D tumor as per the ICRB (International classification of retinoblastoma, Table 2) that present at Rajendra Prasad Centre for Ophthalmic Sciences over first 2 years of the study period

Exclusion Criteria:

* Biomicroscopic evidence of iris neovascularization
* Neovascular glaucoma
* Tumor invasion into the anterior chamber, iris, optic nerve, choroid, or extraocular tissues as documented by clinical, ultrasonographic, and neuroimaging modalities.
* Systemic exclusion criteria include:

  * evidence of systemic metastasis
  * prior chemotherapy
  * prior treatment for retinoblastoma, or
  * inadequate renal or hepatic function

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-04; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Ocular salvage rates in two randomly divided groups of group C and D retinoblastomas, treated with primary chemotherapy protocol using 560mg/m2 carboplatin and 750mg/m2 carboplatin respectively | 1 year

SECONDARY OUTCOMES:
To evaluate the response of subtenon carboplatin injections in cases of group C and D retinoblastomas that fail to respond to primary chemotherapy and local treatment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rachna Meel, MS Ophthal, Principal Investigator — Dr RPC, AIIMS; Supriyo Ghose, MS Ophthal, Study Chair — Prof and HOD, Dr RPC, AIIMS; Sameer Bakhshi, MD Paeds, Study Chair — Associate Prof., IRCH, AIIMS; Neelam Pushker, MD Ophthal, Study Chair — Associate Prof., Dr RPC, AIIMS
Locations (1):
- Dr RPC AIIMS, Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Meel R, Bakhshi S, Pushker N, Vishnubhatla S. Randomized, controlled trial in groups C and D retinoblastoma. Ophthalmology. 2015 Feb;122(2):433-5. doi: 10.1016/j.ophtha.2014.09.013. Epub 2014 Oct 22. No abstract available. PMID 25439612